CLINICAL TRIAL: NCT06443424
Title: Preoperative Assessment of Pediatric Challenging Airway and Endotracheal Tube Sizing Using Point-of-Care Ultrasound Versus Traditional Methods in Elective Surgeries
Brief Title: Assessment of Pediatric Challenging Airway
Status: Not yet recruiting | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Heba Helmy Elshair, assistant lecturer of Anesthesia, Intensive care and PaiN Managment, Zagazig University
Other Study IDs: pocus in pediatric airway
Record Dates: First submitted 2024-05-30; First posted 2024-06-05 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Airway Complication of Anesthesia
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day

INTERVENTIONS:
Device: ultrasound device — usage of ultrasound device in pediatric airway asessment

SUMMARY:
The goal of these Observational study is to learn about pediatric airway the main question to answer is:

1-Is using point-of-care ultrasound provide an easy, early, and accurate preoperative assessment of the challenging pediatric airway and the endotracheal tube sizing more than traditional methods.

ELIGIBILITY:
Inclusion Criteria:

* Patient's parents' consent.
* Age:from one to 4 years old.
* Both sexes (male and female).
* BMI with in (5-85%) of body mass index of the child birth of same age and sex.
* Physical status: American Society of Anesthesiologists (ASA) physical status I and II.
* Type of operation: elective surgery under general anesthesia with endotracheal intubation

Exclusion Criteria:

* Pre-existing airway malformations or pathology like facial or cervical fracture
* Deformity of the airway anatomy [by masses or tumors].
* Pathology of the airway [edema, burn and arthritis].
* Anticipated difficult airway

Ages: 1 Year to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: pediatric population
Sampling Method: Non-Probability Sample
Enrollment: 101 (Estimated)
Dates: Start 2024-07-25 (Estimated); Primary Completion 2025-01-05 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Estimation of tube size using point of care ultrasound compared to age formula in pediatric population | pre induction
  estimate tubal size by ultasound parameters;distance from the skin to the anterior part of the trachea at the hyoid level (ANS-hyoid), The Anterior Neck Soft Tissue Thickness at the level of the vocal Cords. (ANS-VC), The pre - epiglottic space (Pre-E ), the distance from the epiglottis to the mid - point of the distance between the vocal cords (E-VC) , The subglottic transverse diameter and compare with age formula in pediatric

SECONDARY OUTCOMES:
Determine the accuracy of point of care ultrasound in assessing challenging pediatric airway | pre induction
  determine the accuracy of point of care ultrasound in assessing challenging pediatric airway in correlation to Cormack Lehane grading in pediatric patients
Record any obstacles that may interfere with the ultrasound | during opeartion
  ● To record any obstacles that may interfere with the ultrasound assessment such as: acoustic, anatomic , optical illusion artifact.

CONTACTS AND LOCATIONS:
Overall Officials: heba elshair, M.B, B.Ch, Principal Investigator — Anesthesia, Intensive care and Pain Managment Department, Faculty of medicine, Zagazig university
Locations (1):
- Faculty of Medicine, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Background] Santillanes G, Gausche-Hill M. Pediatric airway management. Emerg Med Clin North Am. 2008 Nov;26(4):961-75, ix. doi: 10.1016/j.emc.2008.08.004. PMID 19059095
- [Background] Brambrink AM, Braun U. Airway management in infants and children. Best Pract Res Clin Anaesthesiol. 2005 Dec;19(4):675-97. doi: 10.1016/j.bpa.2005.07.002. PMID 16408541
- [Background] Litman RS, McDonough JM, Marcus CL, Schwartz AR, Ward DS. Upper airway collapsibility in anesthetized children. Anesth Analg. 2006 Mar;102(3):750-4. doi: 10.1213/01.ane.0000197695.24281.df. PMID 16492823
- [Background] Krishna SG, Bryant JF, Tobias JD. Management of the Difficult Airway in the Pediatric Patient. J Pediatr Intensive Care. 2018 Sep;7(3):115-125. doi: 10.1055/s-0038-1624576. Epub 2018 Jan 28. PMID 31073483
- [Background] Mirghassemi A, Soltani AE, Abtahi M. Evaluation of laryngoscopic views and related influencing factors in a pediatric population. Paediatr Anaesth. 2011 Jun;21(6):663-7. doi: 10.1111/j.1460-9592.2011.03555.x. Epub 2011 Mar 14. PMID 21401798
- [Background] Lee SU, Jung JY, Kim DK, Kwak YH, Kwon H, Cho JH, Park JW, Choi YJ. New decision formulas for predicting endotracheal tube depth in children: analysis of neck CT images. Emerg Med J. 2018 May;35(5):303-308. doi: 10.1136/emermed-2017-206795. Epub 2018 Feb 6. PMID 29437848
- [Background] Lin J, Bellinger R, Shedd A, Wolfshohl J, Walker J, Healy J, Taylor J, Chao K, Yen YH, Tzeng CT, Chou EH. Point-of-Care Ultrasound in Airway Evaluation and Management: A Comprehensive Review. Diagnostics (Basel). 2023 Apr 25;13(9):1541. doi: 10.3390/diagnostics13091541. PMID 37174933
- [Background] Pan S, Lin C, Tsui BCH. Neonatal and paediatric point-of-care ultrasound review. Australas J Ultrasound Med. 2022 Oct 13;26(1):46-58. doi: 10.1002/ajum.12322. eCollection 2023 Feb. PMID 36960139
- [Background] Sotoodehnia M, Khodayar M, Jalali A, Momeni M, Safaie A, Abdollahi A. Prediction of difficult laryngoscopy / difficult intubation cases using upper airway ultrasound measurements in emergency department: a prospective observational study. BMC Emerg Med. 2023 Jul 25;23(1):78. doi: 10.1186/s12873-023-00852-4. PMID 37491186
- [Background] Sutagatti JG, Raja R, Kurdi MS. Ultrasonographic Estimation of Endotracheal Tube Size in Paediatric Patients and its Comparison with Physical Indices Based Formulae: A Prospective Study. J Clin Diagn Res. 2017 May;11(5):UC05-UC08. doi: 10.7860/JCDR/2017/25905.9838. Epub 2017 May 1. PMID 28658880